CLINICAL TRIAL: NCT04507581
Title: Evaluation of Atelectasis Formation with Electrical Impedance Tomography During Anesthesia for MRI in Children
Acronym: ATLANTIS
Status: Terminated | Type: Observational
Why Stopped: unsufficient number of partecipants recruited
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Principal Investigator, Thomas Riva, Prof. Dr. med., Insel Gruppe AG, University Hospital Bern
Other Study IDs: 2020-01421
Record Dates: First submitted 2020-08-06; First posted 2020-08-11 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Anesthesia
Keywords: children; electrical impedance tomography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: electrical impedance tomography during anaesthesia — Before induction of the anaesthesia, before the radiological procedure when the induction is terminated, after the termination of the radiological procedure, before transport to the Post anaesthesia Care Unite (PACU), and before the discharge from the PACU after 2 hours of monitoring ventilation distribution changes by thoracic electrical impedance tomography are measured (each measurement will last 1 min). For this, resulting potential differences are measured, and impedance distribution sampled at 30 Hz will be calculated by an automated linearized Newton-Raphson reconstruction algorithm (9). Relative change in poorly ventilated lung regions (silent spaces) and end-expiratory lung impedance (EELI) and measures of ventilation inhomogeneity such as the global inhomogeneity index will be calculated as described previously, using customised software (Matlab R2013a, The MathWorks, Nattick, Massachusetts, USA)(10-12).

SUMMARY:
This study investigates under controlled conditions the variation of poorly ventilated lung units (silent spaces) in children between 1 and 6 years of age measured by electrical impedance tomography during intravenous anaesthesia in a day-hospital setting and before discharge to help further raise safety standards in paediatric anaesthesia

DETAILED DESCRIPTION:
Eligible, children, with parental written informed consent, scheduled for a cerebral magnetic resonance image (MRI) will receive an intravenous anaesthesia using a Propofol infusion of 10 mg/kg/h. At the Bern Children's Hospital all children will be premedicated with Midazolam rectal/oral 0.5 mg/kg or Dexmedetomidine nasal 2 mcg/kg 20 minutes before the beginning of the procedure Eligible children will be prepared for procedure according to the local SOPs of the paediatric anaesthesia departments. Mandatory monitoring will consist of: SpO2, HR, NIBP. An iv-line for drugs injection will be placed.

Induction of anaesthesia: after iv-line placement a bolus of Propofol of 2 mg/kg followed by a continuous infusion of 10 mg/kg/h will be applied. Administration of low-flow oxygen for all children (0.3 l/kg/min) via Microstream® Smart CapnoLine® paediatric cannula (Philips Healthcare, Amsterdam, Netherlands). This cannula allows to measure the etCO2.

In case of extremely agitated child an inhalative induction may be performed. This technique represent the actual standard of care and is not associated with increased risks because of the study.

Before induction of the anaesthesia, before the radiological procedure when the induction is terminated, after the termination of the radiological procedure, before transport to the Post anaesthesia Care Unite (PACU), and before the discharge from the PACU after 2 hours of monitoring ventilation distribution changes by thoracic electrical impedance tomography are measured (each measurement will last 1 min).

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status 1 to 3,
* 1 to 6 years of age with legal guardians providing written informed consent.

Exclusion Criteria:

* Exclusion criteria are necessity to intubate the child,
* contraindication for propofol administration,
* congenital heart or lung disease with oxygen
* dependency and high aspiration risk (requiring rapid sequence induction intubation).

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: We will include paediatric patients undergoing radiological procedures requiring intravenous anaesthesia.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-07-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Changes in poorly ventilated lung areas at 2 Hours after intervention | 2 hours
  Changes in poorly ventilated lung areas (silent spaces) by using electrical impedance tomography (EIT) 2 hours after the end of anaesthesia before discharge at home, which will help quantify the degree of atelectasis

SECONDARY OUTCOMES:
2 min after Anesthesia induction | 2 minutes after the end of anaesthesia induction
  Changes in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT) 2 minutes after the end of induction, before the radiological procedure.
end of the radiological procedure. | 2 minutes after the end of radiological procedure
  Changes in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT) at the end of the radiological procedure
2 minutes after the end of anaesthesia | 2 minutes after the end of anaesthesia, before the transport in Post Anaesthesia Care Unit
  Changes in silent spaces and end-expiratory lung impedance (EELI) by using electrical impedance tomography (EIT) 2 minutes after the end of anaesthesia, before the transport in PACU.
Duration of radiological procedure. | minutes
  Duration of radiological procedure.
Duration of anaesthesia | minutes
  Duration of anaesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Riva, MD, Principal Investigator — University of Bern
Locations (1):
- University Hospital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riva T, Pascolo F, Huber M, Theiler L, Greif R, Disma N, Fuchs A, Berger-Estilita J, Riedel T. Evaluation of atelectasis using electrical impedance tomography during procedural deep sedation for MRI in small children: A prospective observational trial. J Clin Anesth. 2022 May;77:110626. doi: 10.1016/j.jclinane.2021.110626. Epub 2021 Dec 10. PMID 34902800